CLINICAL TRIAL: NCT07060781
Title: Management of Seroma After Posterior Lumbar Spine Decompression
Status: Recruiting | Type: Observational
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ayman Mohamed Basha, Lecturer of Neurosurgery, Faculty of Medicine, KafrElsheikh University, KafrElsheikh, Egypt, Kafrelsheikh University
Other Study IDs: KFSIRB200-645
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Seroma; Lumbar Spine Decompression
MeSH Terms: conditions — Seroma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients undergoing elective posterior lumbar spine decompression.
  Interventions: Procedure: Posterior Lumbar Spine Decompression

INTERVENTIONS:
Procedure: Posterior Lumbar Spine Decompression — Patients undergoing elective posterior lumbar spine decompression.

SUMMARY:
The aim of this study is to evaluate the clinical presentation and management strategies of seroma formation following posterior lumbar spine decompression.

DETAILED DESCRIPTION:
Posterior lumbar spine decompression is a widely employed surgical approach to alleviate neural element compression due to degenerative spinal conditions such as spinal stenosis, spondylolisthesis, and disc herniation. While generally effective in reducing symptoms and improving quality of life, this procedure is not without risk.

Seroma formation, in particular, may follow posterior decompressive surgery or fusion and is thought to arise from the accumulation of lymphatic or serous fluid in the dead space created by tissue dissection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both sexes.
* Patients undergoing elective posterior lumbar spine decompression.

Exclusion Criteria:

* History of previous lumbar spine surgery.
* Active spinal infection, trauma, or malignancy.
* Severe medical comorbidities that contraindicate surgery or influence wound healing (e.g., uncontrolled diabetes, immunosuppression, severe cardiovascular disease).
* Patients unfit for general anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study will be conducted on 50 adult patients undergoing posterior lumbar spine decompression surgery at Kafr Elsheikh University Hospitals. Approval from the Medical Sciences Ethics Committee of Kafr Elsheikh Faculty of Medicine will be taken. Written informed consent will be obtained from all participants before enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-07-19 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of seroma | 6 months postoperatively
  Incidence of seroma formation following posterior lumbar spine decompression will be recorded during hospitalization and at scheduled postoperative follow-up visits at 2 weeks, 6 weeks, 3 months, and 6 months.

SECONDARY OUTCOMES:
Number of aspirations required | 6 months postoperatively
  Number of aspirations required will be recorded.
Seroma recurrence rate | 6 months postoperatively
  Seroma recurrence rate will be recorded.
Association with patient risk factor | 6 months postoperatively
  Association with patient risk factor will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.